CLINICAL TRIAL: NCT06426433
Title: Investigation of The Effects of Proprioceptive Exercise Training on Motor Performance Parameters in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Cigdem Ayhan, Professor Doctor of Physical Therapy and Rehabilitation Faculty, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-94603339-604.01.02-268134
Record Dates: First submitted 2024-05-15; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Exercise; Proprioception; Wrist Injuries
Keywords: Wrist; Proprioception
MeSH Terms: conditions — Motor Activity; Wrist Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wrist Proprioceptive Exercises and General Upper Extremity Exercises (Other): Wrist Proprioceptive Exercises are neuromuscular exercises for wrist stabilization and control.
  Interventions: Other: Proprioceptive Exercises; Other: Upper Extremity Exercises
- General Upper Extremity Exercises (Other): These exercises are traditional rehabilitation exercises.
  Interventions: Other: Upper Extremity Exercises

INTERVENTIONS:
Other: Proprioceptive Exercises — In our study, participants were divided into two different exercise groups, starting with the same warm-up exercise program, and a 6-week exercise training program was implemented. To reduce the potential error resulting from daily life activities, exercise training was given to the non-dominant side of the participants. Proprioceptive exercises aim to restore muscle balances, unconscious joint control with reactive muscle activations and feedforward joint control.
  Arms: Wrist Proprioceptive Exercises and General Upper Extremity Exercises
Other: Upper Extremity Exercises — In our study, participants were divided into two different exercise groups, starting with the same warm-up exercise program, and a 6-week exercise training program was implemented. To reduce the potential error resulting from daily life activities, exercise training was given to the non-dominant side of the participants. Upper extremity exercises are traditional rehabilitation exercises for strength, endurance and range of motion.

SUMMARY:
This study was conducted to investigate the effect of two different exercise protocols applied to healthy individuals on motor performance parameters. Forty-one healthy participants were included in the study. Participants were divided into 2 groups (wrist proprioceptive exercise group, general exercise group) and attended exercise training targeting the hand and wrist for a total of 6 weeks. Before and after the exercises, sociodemographic evaluation, Quick Disability of Arm Shoulder and Hand questionnaire, pain assessment, grip strength measurement, weight transfer tolerance test, wrist joint position sense, Nelson hand reaction test, upper extremity Y balance test, lateral grip and tripod grip measurements, manual muscle testing, and surface electromyography analysis were evaluated in both groups.

DETAILED DESCRIPTION:
Healthy volunteers who met the inclusion criteria were included in the study upon agreement to participate. The participants were divided into two groups. One group received 6 weeks of general upper extremity exercises along with proprioceptive exercise training. The proprioceptive exercise training consisted of a 10-minute warm-up period including active and passive upper extremity exercises followed by 30 minutes of proprioceptive exercises. The exercise program progressed weekly, and exercises were performed in standardized positions. To ensure adherence to the exercises, they were recorded on video and sent to participants' phones. The second group performed general upper extremity exercises for 6 weeks. The reason for creating the second group was to eliminate the time-dependent effect of changes in electromyographic activation levels of muscles. Additionally, the bilateral effects of unilateral upper extremity exercise training are observed. Comparing the electromyographic activities of untrained healthy individuals at the end of the treatment may enhance the quality of data interpretation. However, other factors that increase the risk of error in evaluating distal motor performance of the upper extremity were also considered in our study. It is expected that the motor performance of the dominant side will be greater than that of the non-dominant side. However, the non-dominant side is more frequently used in daily activities, resulting in a higher frequency and intensity of daily life activities being loaded onto the dominant side. To reduce the potential error resulting from daily life activities, exercise training was given to the non-dominant side of the healthy individuals participating in our study. Detailed evaluations were performed on the individuals participating in the study, as described below. Evaluations were conducted twice, before starting the exercise program and after the 6-week exercise program.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18 and 30
* To be willing to participate in the study
* To have cognitive abilities to understand the tasks required in the study.

Exclusion Criteria:

* Experiencing acute/chronic bilateral or unilateral upper extremity pain
* Having neurological and/or rheumatological diseases
* Chronic medication usage
* Regular smoking/alcohol consumption currently or in the past
* Taking cortisone orally or via injection
* Suffering from upper extremity musculoskeletal injuries in the past year
* Undergoing upper extremity surgery
* Having a body mass index greater than 24.9 kg/m2
* Scoring above 6 on the Beighton hypermobility score
* Engaging in regular exercises involving the upper extremities
* History of autoimmune and/or rheumatic diseases
* Regular use of anti-inflammatory medications, etc.
* Having cardiovascular disease and diabetes

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Surface Electromyography | Within the week before starting the exercise and within the week after finishing the exercise
  Measurement of wrist muscles activation levels

SECONDARY OUTCOMES:
Grip Force | Within the week before starting the exercise and within the week after finishing the exercise
  Measurement of hand grip force
Weight Bearing Tolerance Test | Within the week before starting the exercise and within the week after finishing the exercise
  Measurement of weight bearing capacity of healthy wrist
Joint Position Sense | Within the week before starting the exercise and within the week after finishing the exercise
  Measurement of position senses for 4 wrist range of motion directions
Reaction time | Within the week before starting the exercise and within the week after finishing the exercise
  Measurement of Nelson hand reaction time
Upper extremity y balance test | Within the week before starting the exercise and within the week after finishing the exercise
  Measurement of upper extremity balance and mobility
Tripod grip | Within the week before starting the exercise and within the week after finishing the exercise
  Measurement of tripod hand grip force
Lateral grip | Within the week before starting the exercise and within the week after finishing the exercise
  Measurement of lateral hand grip force
Manual muscle test | Within the week before starting the exercise and within the week after finishing the exercise
  Measurement of manual muscle dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Semiha Tomiris Erzincanlı, MSc Student, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)